CLINICAL TRIAL: NCT01421277
Title: Migraine Attack Study of Treatment, Efficacy and Resource Use (MASTER) - McKesson Substudy (MK-0974-076)
Brief Title: Study of Treatment Used for Migraine Headaches (MK-0974-076)
Acronym: MASTER
Status: Terminated | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0974-076
Record Dates: First submitted 2011-07-28; First posted 2011-08-22 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Participants Enrolled in Protocol Version (V)1.1: Participants with physician-diagnosed migraine with or without aura who are treatment-naive to triptans, who received their first prescription for a triptan and took at least one dose within 6 months prior to being included in Protocol V1.1 of this study.
  Interventions: Drug: Statin Therapy
- Participants Enrolled in Protocol V2: Participants with physician-diagnosed migraine with or without aura who are treatment-naive to triptans, who received their first prescription for a triptan and took at least one dose within 6 months prior to being included in Protocol V2 of this study.
  Interventions: Drug: Statin Therapy

INTERVENTIONS:
Drug: Statin Therapy — Investigator's choice of any statin.

SUMMARY:
This study will describe the reasons for triptan utilization patterns (continuation and discontinuation) in triptan-naïve participants and assess the stability of treatment utilization patterns over time according to standard medical guidelines or clinical practice standards of the investigating physician.

DETAILED DESCRIPTION:
After study start, the Protocol was amended to clarifiy that the first triptan prescription must have been received by the participant within a time window of 3 months (± 2 weeks) prior to the participant being identified by the Investigator, and could be enrolled into the study within 6 months of taking the prescribed triptan medication for the first time and that use of a sample triptan would not disqualify a participant as long as the sample was of the same triptan that was eventually prescribed.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years of age in the United States at the time of consent
* Physician-diagnosed migraine with or without aura
* At least two and up to a maximum of 8 moderate to severe migraine attacks during the 30 days prior to screening
* Initial triptan prescription 3 months (± 2 weeks) prior to being identified as eligible for this study, and triptan-naïve before that initial prescription
* Used triptan medication at least once within 6 months prior to the date of informed consent for screening
* Internet access and able to complete online surveys via electronic data entry

Exclusion criteria:

* Treated with triptans prior to this study
* In active litigation and compensation issues including disability dispute cases with a Government agency
* Participation in a clinical trial within the last 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with physician-diagnosed migraine (with or without aura) who have had at least two, but not more than 8 moderate to severe migraines during the 30 days prior to screening. Participants must have received a triptan prescription 3 months (± 2 weeks) prior to being identified by the physician, must have been triptan-naïve prior to that initial prescription, and must have taken triptan medication at least once within 6 months prior to the date of informed consent for screening.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2011-05-19 (Actual); Primary Completion 2012-03-23 (Actual); Study Completion 2012-03-23 (Actual)

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=0974-076&kw=0974-076&tab=access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 216 of the 806 screened participants were eligible for the study and were invited to participate in the online survey.
Period: Overall Study
Arm/Group | Participants Enrolled in Protocol Version (V)1.1 | Participants Enrolled in Protocol V2
Started | 25 | 191
Completed | 25 (Completed the online survey for at least one migraine attack.) | 99 (Completed the online survey for at least one migraine attack.)
Not Completed | 0 | 92
Not completed — Lack of qualifying event | 0 | 61
Not completed — Incomplete baseline data | 0 | 31

BASELINE CHARACTERISTICS:
Population: All eligible particpants. 2 participants did not specify gender in the online questionnaire.
Groups:
- Participants Enrolled in Protocol Version V1.1: Participants with physician-diagnosed migraine with or without aura who are treatment-naive to triptans, who received their first prescription for a triptan and took at least one dose within 6 months prior to being included in Protocol V1.1 of this study.
- Total: Total of all reporting groups
Arm/Group | Participants Enrolled in Protocol Version V1.1 | Participants Enrolled in Protocol V2 | Total
Number analyzed (Participants) | 25 | 191 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.0 (15.77) | 39.8 (13.39) | 39.9 (13.65)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 20 | 157 | 177
  Male | 5 | 32 | 37
  Not reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Using a Triptan for Migraine Attacks
Description: Participants reported information online. For this measure, the number of participants who used at least one dose of any newly prescribed triptan for the first time in response to a migraine attack were counted.
Time Frame: Up to 3 months
Population: All screened participants who were fully eligible for the study.
Measure: Number; unit: Number of participants
Arm/Group | Participants Enrolled in Protocol Version V1.1 | Participants Enrolled in Protocol V2
Number analyzed (Participants) | 25 | 191
Number of participants | 25 | 191

2. Primary Outcome: Number of Participants Continuing Triptan Therapy
Description: Participants reported information online. For this measure, the number of participants who continued to use a triptan after the first migraine attack were counted; switching from one triptan to another was considered continued use.
Time Frame: Up to 3 monoths
Population: All screened participants who were fully eligible for the study.
Measure: Number; unit: Number of participants
Arm/Group | Participants Enrolled in Protocol Version V1.1 | Participants Enrolled in Protocol V2
Number analyzed (Participants) | 25 | 191
Number of participants | 25 | 174

3. Primary Outcome: Main Reason for Stopping Triptan Use
Time Frame: Up to 3 months
Population: All screened participants who were fully eligible for the study.
Measure: Number; unit: Number of partiicpants
Arm/Group | Participants Enrolled in Protocol Version V1.1 | Participants Enrolled in Protocol V2
Number analyzed (Participants) | 25 | 191
Number of partiicpants
  Other medications worked better | 0 | 2
  Side effects of triptan | 0 | 5
  Insurance stopped covering cost | 0 | 2
  Physician or health care provider decision | 0 | 1
  Triptan did not work | 0 | 7

ADVERSE EVENTS:
Description: Adverse events were not collected for this study.
Arm/Group | Participants Enrolled in Protocol Version V1.1 | Participants Enrolled in Protocol V2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.